CLINICAL TRIAL: NCT05338307
Title: Preliminary Investigation of β-hydroxybutyrate Supplementation in Colorectal Cancer
Brief Title: Preliminary Investigation of β-hydroxybutyrate Supplementation in Colorectal Cancer Prevention
Acronym: BHB-CRC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UPCC 01222; IRB 850567 (Other: University of Pennsylvania Abramson Cancer Center)
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — beta-hydroxybutyrate-1,3-butanediol monoester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BHB supplementation (Experimental): Study participants will be taking 35mL of HVMN Ketone-IQ by mouth three times daily, with each dose containing 10 grams of R-1,3-Butanediol, for a total of 4 weeks.
  Interventions: Dietary Supplement: R-1,3-Butanediol

INTERVENTIONS:
Dietary Supplement: R-1,3-Butanediol — Study participants will be taking 35mL of HVMN Ketone-IQ by mouth three times daily, with each dose containing 10 grams of R-1,3-Butanediol.

SUMMARY:
The aim of this study is to assess the feasibility of beta-hydroxybutyrate (BHB) supplementation in individuals who are undergoing a standard-of-care colonoscopy or flexible sigmoidoscopy.

DETAILED DESCRIPTION:
The aim of this study is to assess the feasibility of β-hydroxybutyrate (BHB) supplementation in individuals who are undergoing a standard-of-care colonoscopy or flexible sigmoidoscopy in order to determine whether BHB supplementation is safe and tolerable. Additionally, this study will determine whether BHB supplementations increases serum BHB levels, and leads to transcription and protein expression changes in the colonic mucosa. BHB supplementation will be performed through oral administration of HVMN Ketone-IQ, a commercially available BHB supplement, with an active ingredient of R-1,3-Butanediol, which gets converted to BHB.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Scheduled for a colonoscopy or flexible sigmoidoscopy as part of the patient's standard care
* Can provide informed consent

Exclusion Criteria:

* Subject is pregnant, a prisoner, or is under 18 years of age
* Patient is not able to undergo colonoscopy or flexible sigmoidoscopy
* Prior total proctocolectomy
* History of inflammatory bowel disease
* History of diabetes mellitus and are currently on medical diabetes therapy
* History of chronic kidney disease with an eGFR < 60 mL/min/1.73m2
* Cancer diagnosis where the subject is receiving active therapy
* Use of either a ketogenic diet or intermittent fasting (defined as a fasting period of 16 hours or more per day that is not associated with a medical procedure) during the 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine whether oral BHB supplementation is safe and tolerable | Through study completion, which will be approximately 2 years
  Assessment of patient tolerance of BHB supplements through weekly monitoring of side effects and/or intolerances and patient compliance. We will monitor the percentage of individuals who continue through Visit 2, and the percentage continuing through Visit 3, as well as the compliance with taking the BHB supplement.

SECONDARY OUTCOMES:
Determine whether oral BHB supplementations increases serum BHB levels | Through study completion, which will be approximately 2 years
  Assessment of fasting serum BHB levels before, during, and after BHB supplementation to determine if BHB supplementation appreciably increases serum BHB levels.
Investigate whether oral BHB supplementation leads to transcription and protein expression changes in the colonic mucosa | Through study completion, which will be approximately 2 years
  Comparison of both transcription and protein changes in the colonic mucosa from mucosal biopsies before and after BHB supplementation to determine if BHB supplementation is having measurable effects on the colonic mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Bryson W Katona, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No